CLINICAL TRIAL: NCT07394829
Title: Evaluation of the Effects of Different Compression Pressure Levels on Lower Extremity Peripheral Circulation in the Postoperative Period: A Pilot Study
Brief Title: Effects of Different Compression Pressure Levels on Peripheral Circulation After Surgery
Acronym: COMP-PILOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Agri Ibrahim Cecen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AICU-COMP-POSTOP-2026
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Circulatory Changes; Peripheral Vascular Diseases; Venous Insufficiency of Leg
Keywords: Elastic compression; Compression pressure; Postoperative care; Peripheral perfusion index; Lower extremity circulation; Pilot study
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: All participants will receive sequential compression pressure levels applied in a single group design, with repeated measurements at each pressure level within the same participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential Compression Pressure Intervention (Experimental): All participants will receive sequential lower extremity compression at three predefined pressure levels (30 mmHg, 45 mmHg, and 60 mmHg) applied to the calf region during the early postoperative period, with repeated measurements at each pressure level within the same participant.
  Interventions: Device: Pressure-Controlled Compression Device

INTERVENTIONS:
Device: Pressure-Controlled Compression Device — A pressure-controlled compression device will be applied to the calf region to deliver sequential compression at three predefined pressure levels: low (30 mmHg), moderate (45 mmHg), and high (60 mmHg). Each pressure level will be applied for a fixed duration with rest periods between applications to allow peripheral circulation to return to baseline. Compression will be performed in the supine position during the early postoperative period.

SUMMARY:
After surgery, elastic compression is commonly used on the legs to support blood circulation and reduce the risk of complications such as swelling and venous thromboembolism. In clinical practice, compression is usually applied at fixed pressure levels, although individual patients may respond differently depending on their circulation and tissue tolerance.

The purpose of this pilot study is to evaluate how different compression pressure levels affect peripheral circulation in adult patients during the early postoperative period. Participants will receive three different levels of leg compression applied sequentially under controlled conditions. Peripheral circulation will be assessed using non-invasive methods, including photoplethysmography and peripheral perfusion index measurements.

The findings of this study are expected to provide preliminary evidence on individual circulatory responses to different compression pressures and to support the development of more personalized postoperative compression strategies in future clinical practice.

DETAILED DESCRIPTION:
Elastic compression therapy is a standard component of postoperative care aimed at improving venous return, reducing lower extremity edema, and supporting peripheral circulation. Despite its widespread use, compression is commonly applied using fixed pressure levels without systematic consideration of individual circulatory responses. This may result in suboptimal effectiveness or discomfort in some patients.

This study is designed as a prospective, single-center pilot interventional study to investigate the effects of different compression pressure levels on lower extremity peripheral circulation in adult postoperative patients. The study will be conducted in surgical wards of Ağrı Training and Research Hospital. Adult patients who have undergone elective surgery and are hemodynamically stable will be enrolled during the early postoperative period.

Each participant will receive three sequential compression pressure levels applied to the calf region using a pressure-controlled compression device. The predefined pressure levels are low (30 mmHg), moderate (45 mmHg), and high (60 mmHg). Compression will be applied in a supine position following a standardized rest period. Each pressure level will be maintained for a fixed duration, with adequate rest intervals between applications to allow circulation to return to baseline.

Peripheral circulation will be assessed at baseline and after each compression level using non-invasive measurement techniques. The primary outcome measures include peripheral perfusion index and venous filling time assessed by photoplethysmography. Secondary outcome measures include lower extremity edema, skin surface temperature, and patient-reported comfort assessed using a visual analog scale. Safety and tolerability will be monitored throughout the study, and compression will be discontinued immediately if any discomfort or adverse effects occur.

As a pilot study, the planned sample size is limited and no formal power calculation has been performed. The primary objective is to generate preliminary data on circulatory responses to different compression pressures and to evaluate the feasibility of the study protocol. The results are intended to inform the design of future larger-scale clinical trials and contribute to evidence-based, individualized postoperative compression practices.

The study will be conducted in accordance with the Declaration of Helsinki. Ethics committee approval was obtained prior to study initiation, and written informed consent will be obtained from all participants before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Undergoing elective surgery
* In the early postoperative period at the time of assessment
* Hemodynamically stable
* Intact skin on the lower extremities at the planned compression sites
* Able to understand the study procedures
* Willing and able to provide written informed consent

Exclusion Criteria:

* Peripheral arterial disease or clinically significant arterial insufficiency
* Current or previous diagnosis of deep vein thrombosis or venous thromboembolism
* Known peripheral neuropathy or sensory impairment affecting the lower extremities
* Open wounds, active infection, or dermatological conditions on the lower extremities
* Severe edema requiring therapeutic intervention beyond standard postoperative care
* Inability to tolerate compression therapy due to pain or discomfort
* Pregnancy
* Participation in another interventional clinical study during the same hospitalization period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Peripheral Perfusion Index (PPI) | Baseline (T0) and during sequential compression applications (T1-T3) within the first 48 hours after surgery
  Peripheral Perfusion Index (PPI) will be measured as a dimensionless numerical value using a non-invasive photoplethysmography-based monitoring device. PPI represents the ratio of pulsatile to non-pulsatile blood flow and serves as an objective indicator of peripheral microcirculatory perfusion.
  Measurements will be obtained at four predefined time points: baseline before compression (T0), after application of 30 mmHg compression (T1), after application of 45 mmHg compression (T2), and after application of 60 mmHg compression (T3). All measurements will be performed in the supine position following a standardized rest period of at least 10 minutes.
Venous Filling Time Measured by Photoplethysmography (seconds) | Baseline (T0) and during sequential compression applications (T1-T3) within the first 48 hours after surgery
  Venous filling time will be measured in seconds (s) using non-invasive photoplethysmography to assess venous hemodynamic response of the lower extremity. Venous filling time reflects the rate of venous refilling following compression release.
  Measurements will be recorded at baseline (T0) and after each compression pressure level: 30 mmHg (T1), 45 mmHg (T2), and 60 mmHg (T3), using standardized sensor placement at the calf region in the supine position.
  .

SECONDARY OUTCOMES:
Lower Extremity Edema (Circumference Measurement, cm) | Baseline (T0) and during sequential compression applications (T1-T3) within the first 48 hours after surgery
  Lower extremity edema will be assessed by circumferential tape measurements (centimeters) at standardized anatomical landmarks, including the ankle (malleolar level) and calf (maximum circumference), at baseline and after each compression pressure level.
Skin Surface Temperature (°C) | Baseline (T0) and during sequential compression applications (T1-T3) within the first 48 hours after surgery
  Skin surface temperature of the lower extremity will be measured in degrees Celsius (°C) using non-invasive thermal sensors to assess peripheral thermal response associated with different compression pressure levels.
Patient Comfort Assessed by Visual Analog Scale (VAS, 0-10) | Baseline (T0) and during sequential compression applications (T1-T3) within the first 48 hours after surgery
  Patient comfort and tolerance will be assessed using a Visual Analog Scale (VAS) ranging from 0 (no discomfort) to 10 (maximum discomfort). The VAS score will be recorded after each compression pressure level to evaluate subjective comfort during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Training and Research Hospital, Ağrı, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the pilot nature of the study, the small sample size, and the single-center design. The collected data include detailed physiological measurements that could potentially increase the risk of participant re-identification. Aggregate and de-identified results will be reported in scientific publications in accordance with ethical approval and data protection regulations.

REFERENCES:
- [Background] Furukawa H. Furukawa H: Some problems in esophageal reconstruction regarding the tissue respiration of the digestive tract. Nihon Geka Hokan. 1967 Sep 1;36(5):565-87. No abstract available. PMID 4229808
- [Background] Kageyama M, Nakatsuka K, Miyake Y. [A case of congenital retinoschisis with unexpected appearance and spontaneous regression]. Nippon Ganka Gakkai Zasshi. 1997 Aug;101(8):698-702. Japanese. PMID 9284627
- [Background] Reynolds JD, Hiles DA, Johnson BL, Biglan AW. Hyperplastic persistent pupillary membrane--surgical management. J Pediatr Ophthalmol Strabismus. 1983 Jul-Aug;20(4):149-52. doi: 10.3928/0191-3913-19830701-06. PMID 6886954
- [Background] Sun X, He H, Xu M, Long Y. Peripheral perfusion index of pulse oximetry in adult patients: a narrative review. Eur J Med Res. 2024 Sep 11;29(1):457. doi: 10.1186/s40001-024-02048-3. PMID 39261939
- [Background] Bode J, Benham C, Ernst E, Knopp A, Marschalek R, Strick R, Strissel P. Fatal connections: when DNA ends meet on the nuclear matrix. J Cell Biochem Suppl. 2000;Suppl 35:3-22. doi: 10.1002/1097-4644(2000)79:35+3.0.co;2-9. PMID 11389527